CLINICAL TRIAL: NCT06741241
Title: Effectiveness of an EHealth Intervention for Uptake of Cervical Cancer Screening in Hispanic Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida A&M University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2180042-1; 2U54MD007582-39 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the eHealth promotora intervention where they will participate in a group education session of cervical cancer screening or a control group where they will participate in a group education session on healthy nutrition.
Who Masked: Participant
Masking Description: Participants will complete surveys and receive virtual education sessions and not know if they are in control arm or intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eHealth Promotora (Experimental): Intervention arm participants will participate in a eHealth promotora group education session to receive a presentation on cervical cancer screening education, view an educational video, and complete baseline and 6-month follow-up surveys.
  Interventions: Behavioral: eHealth Promotora
- eHealth Healthy Nutrition (Active Comparator): Control group participants will participate in an eHealth group education session to receive a presentation on healthy nutrition information, view an educational video, and complete baseline and 6-month surveys.
  Interventions: Behavioral: eHealth Healthy Nutrition

INTERVENTIONS:
Behavioral: eHealth Promotora — Intervention participants attend an eHealth promotora-delivered educational session. Activities include an icebreaker, the completion of a baseline survey, an introduction to cervical cancer using a video and slide presentation, a cervical cancer knowledge pretest/posttest, and a dialogue activity to explore possible barriers and solutions to health care access. Main topics included in the slide presentation are: female anatomy; cervical cancer etiology and disease progression by stage; cancer prevention including diet, exercise, safe sex, cancer screening; human papillomavirus (HPV) vaccine recommendations; Pap test preparations, procedure, screening interval; and information about where to receive a Pap test and seek more information about cervical cancer.
  Arms: eHealth Promotora
Behavioral: eHealth Healthy Nutrition — Control group participants attend an eHealth educational session on healthy nutrition. Activities include an icebreaker, the completion of a baseline survey, an introduction to healthy eating using a video and a slide presentation, a cervical cancer knowledge pretest/posttest, and a dialogue activity to explore benefits and challenges to healthy eating.
  Arms: eHealth Healthy Nutrition

SUMMARY:
This study will test the effectiveness of an eHealth promotora (lay health advisor) outreach strategy to increase cervical cancer screening in Hispanic women. The investigators will recruit 160 Hispanic women ages 21-65 who are not up to date with cervical cancer screening or have never been screened, with the goal to evaluate screening knowledge, behavior, and intervention effects on cervical cancer screening outcomes. The study will utilize a two-arm, cluster randomized trial design, and participants will be randomly assigned to the cervical cancer education intervention or a nutrition education control group. The cervical cancer education arm will utilize a promotora to deliver an educational session virtually to encourage cervical cancer screening and receive a resource list for screening sites. The control group will participate in an educational session virtually about the importance of healthy nutrition. The primary study outcome is receipt of cervical cancer screening measured six months following receiving the intervention. The secondary outcomes will include cervical cancer screening knowledge and self-efficacy (confidence to receive cervical cancer screening). The research objective is to test the eHealth promotora intervention effectiveness for promoting cervical cancer screening in an under-screened Hispanic population.

ELIGIBILITY:
Inclusion Criteria:

1. between the age of 21 and 65 years
2. identify as Hispanic
3. not up-to-date with cervical cancer screening [never screened or last Pap test ≥ 3 years - based on U.S. Preventive Services Task Force guidelines]
4. have no history of cervical cancer
5. have not had a hysterectomy.

Exclusion Criteria:

1. under the age of 21 or over the age of 65 years
2. do not identify as Hispanic
3. up-to-date with cervical cancer screening [last Pap test < 3 years - based on U.S. Preventive Services Task Force guidelines]
4. history of cervical cancer
5. have had a hysterectomy.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Cervical cancer screening uptake | 6 months
  Proportion of participants who complete cervical cancer screening determined by cervical cancer screening measure which asks about the last Pap test completed confirmed by chart review if possible.

SECONDARY OUTCOMES:
Cervical cancer screening self-efficacy | 6 months
  The 10-item cervical cancer screening self-efficacy scale is scored on a 5-item Likert scale ranging from 1 (very unsure) to 5 (very sure) (α = 0.88). Questions include asking participants to rate their confidence in having a discussion with their doctor about the Pap test, scheduling and keeping appointments, getting a Pap test despite being worried about pain, and overcoming embarrassment.
Cervical cancer knowledge | 6 months
  A 15-item cervical cancer knowledge instrument measures educational content of the intervention with 10 True/False questions and 5 multiple choice questions to produce a knowledge score ranging from 0 to 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida A&M University, Tallahassee, Florida, United States